CLINICAL TRIAL: NCT01833000
Title: Assessment of Splanchnic Oxygenation and Circulation in Neonates at Risk for Necrotizing Enterocolitis Using NIRS and Doppler
Brief Title: NIRS and Doppler to Predict NEC in Risk Neonates
Acronym: NeoNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9048
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Necrotizing Enterolitis
Keywords: rectal bleeding; necrotizing enterolitis; splanchnic oxygenation; mesenteric doppler
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- newborn suspected to suffer from necrotizing enterolitis (Other): Cerebral and splanchnic ear infrared spectroscopy (NIRS) and mesenteric Doppler
  Interventions: Device: Cerebral and splanchnic ear infrared spectroscopy (NIRS) and mesenteric Doppler

INTERVENTIONS:
Device: Cerebral and splanchnic ear infrared spectroscopy (NIRS) and mesenteric Doppler

SUMMARY:
The main objective is to evaluate the interest of cerebro-splanchnic oxygenation ratio (CSOR) for early diagnosis of necrotizing enterocolitis (NEC) in neonates with rectal bleeding and/or abdominal distension. CSOR will be determined using near infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* less than 28 days neonates hospitalised in neonatology care unit presenting rectal bledding and/or abdominal distension
* signed authorization by the parents (consent form)

Exclusion Criteria:

* - cutaneous lesions in the regions of monitoring
* emergency for NEC

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Cerebro-splanchnic oxygenation ratio | up to 48h
  NIRS assessment

SECONDARY OUTCOMES:
Mesenteric Doppler flow | up to 48h

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Cambonie, MD,PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France